CLINICAL TRIAL: NCT03058705
Title: Pilot Study: Assessing Near Infrared Fluorescence Imaging Medical Technology for the Detection of Bladder Cancer
Brief Title: Near Infrared Fluorescence Imaging for Bladder Cancer Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Messing (Other)
Collaborators: Imagin Medical (Unknown)
Responsible Party: Sponsor-Investigator, Edward Messing, Principal Investigator, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 66682
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hexaminolevinulate HCL with Near Infrared Fluorescence (NIRF) (Experimental): During the transurethral resection of the bladder procedure, the bladder will initially be examined in a systematic meridian fashion. Suspicious tumors identified by white light only, NIRF only, and both will be identified. If intense fluorescence is observed in the initial patient(s) at 10 min, dwell duration will be reduced to 5 min for the next patient(s); if abundant fluorescence is detected there as well, dwell duration will be shortened again to 2.5 min. At least three patients will be studied at each duration to document intense fluorescence before proceeding to shorter instillation durations in subsequent patients.
  Interventions: Drug: Hexaminolevulinate HCL; Device: Near Infrared Fluorescence (NIRF)

INTERVENTIONS:
Drug: Hexaminolevulinate HCL — Intravesical instillation of 100 mg hexaminolevulinate HCL will be performed via foley catheter at the initiation of the procedure. Although NIRF is more sensitive than bluelight cystoscopy, the current FDA approved dose will be used. Hexaminolevulinate has a favorable safety profile at this dose.
Device: Near Infrared Fluorescence (NIRF) — NIRF is a highly sensitive multi-spectral imaging modality that speeds the detection of bladder cancer fluorescence after infusion of hexaminolevinulate.

SUMMARY:
The primary outcome of this study is to determine the minimal dwell time needed for adequate detection of hexaminolevinulate HCL avid tumors using protoporphyrin IX (PpIX) near infrared fluorescence (NIRF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bladder mass on office cystoscopy suspicious for malignancy, either newly diagnosed or a recurrent tumor.
* Planned transurethral resection of bladder tumor in the operating room.
* Ability to give informed consent.
* Willing to spend time for the study
* Men or women (age 18 or older)
* Any racial or ethnic origin

Exclusion Criteria:

* Pregnancy
* Nursing mother
* Diagnosis of porphyria
* Gross hematuria
* BCG immunotherapy or intravesical chemotherapy within the past 90 days
* Known hypersensitivity to hexaminolevulinate or any derivative of aminolevulinic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Messing, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Hexaminolevinulate HCL With Near Infrared Fluorescence (NIRF): Patients with possible bladder cancer to be evaluated using near infrared fluorescence imaging (NIRF) device.
  Hexaminolevulinate HCL: Intravesical instillation of 100 mg hexaminolevulinate HCL will be performed via foley catheter at the initiation of the procedure. Although NIRF is more sensitive than bluelight cystoscopy, the current FDA approved dose will be used. Hexaminolevulinate has a favorable safety profile at this dose.
Period: Overall Study
Arm/Group | Hexaminolevinulate HCL With Near Infrared Fluorescence (NIRF)
Started | 10
Completed | 6
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hexaminolevinulate HCL With Near Infrared Fluorescence (NIRF)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Minimal Dwell Time
Description: The minimum time needed to observe the tumors during transurethral resection of bladder tumor (TURBT).
Time Frame: Day 1
Population: Dwell time was not collected on any participant due to failure to visual fluorescence in the subjects.
Arm/Group | Hexaminolevinulate HCL With Near Infrared Fluorescence (NIRF)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Hexaminolevinulate HCL With Near Infrared Fluorescence (NIRF)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03058705/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03058705/ICF_001.pdf